CLINICAL TRIAL: NCT07221461
Title: Prospective, Single Center, Open-label Study Assessing Impact of Microdroplet Hyaluronic Acid Filler on Skin Quality and Biomarkers in Patients on Glucagon-like Peptide-1 Agonists
Brief Title: Assess Impact of Microdroplet Hyaluronic Acid Filler on Skin Quality in Patients on Glucagon-like Peptide-1 Agonists
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Skinvive GLP1 agonist
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Wrinkle
Keywords: skin laxity; fine lines; dull skin; uneven skin tone
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: All subjects (16 GLP1 and 8 non-GLP1) will receive one treatment with microdroplet hyaluronic acid filler (SKINVIVE™, JUVÉDERM®, Irvine, CA) to the cheeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- GLP1 Patients (Active Comparator): 16 participants who have been on a stable dose of GLP-1 agonist medication for at least the last 6 months will receive one treatment with microdroplet hyaluronic acid filler (SKINVIVE™, JUVÉDERM®, Irvine, CA) to the cheeks.
  Interventions: Device: Skinvive
- NON GLP1 Patients (Experimental): 8 participants who are GLP1 naive will receive one treatment with microdroplet hyaluronic acid filler (SKINVIVE™, JUVÉDERM®, Irvine, CA) to the cheeks.
  Interventions: Device: Skinvive

INTERVENTIONS:
Device: Skinvive — 16 GLP1 subjects treated with Skinvive to their cheeks for skin quality will be compared to 8 NON-GLP1 subjects treated with Skinvive for skin quality.

SUMMARY:
Clinical trial to assess the effect of microdroplet hyaluronic acid filler to the cheek skin (SKINVIVE™, JUVÉDERM®, Irvine, CA) on skin quality in patients undergoing medical weight loss with GLP-1 therapy.

DETAILED DESCRIPTION:
24 patients total (16 GLP1 and 8 non-GLP1) will receive one treatment with microdroplet hyaluronic acid filler (SKINVIVE™, JUVÉDERM®, Irvine, CA) to the cheeks, either at the beginning of the study or at the end. Patients will return for follow up visits at day 30, day 60 and and day 70, where they will undergo standardized 2D photography, VISIA photography and assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women aged 25-50 years.
2. Fitzpatrick skin types I-VI.
3. Current treatment with a stable dose of GLP-1 agonist medication for at least the last 6 months, for 16 of the enrolled subjects. Remaining 8 subjects should not be taking or have a history of taking a GLP-1 agonist therapy in the last year.
4. Presence of moderate skin changes (as defined by Modified Griffiths' Scale, with an average score of 4-6) in the following criteria: skin radiance/brightness, skin elasticity, tone evenness, skin firmness, fine lines, global wrinkles, and skin smoothness (tactile and visual).
5. Participants must maintain a stable weight, defined as no greater than a 10% weight change from screening/baseline and throughout the study.
6. Participants must have a body mass index (BMI) of 27 or less.
7. Must be willing to sign a photography release and ICF, and complete the entire course of the study.
8. Participant must agree to maintaining the same skincare routine they are currently using throughout the study period.
9. Subjects in good general health based on investigator's judgment and medical history.
10. Negative urine pregnancy test result at the time of study entry (if applicable).
11. Females of childbearing potential must be willing to use an acceptable method of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

    1. 1. Acceptable methods of birth control are: oral contraceptive pill, injections, implants, patches, vaginal rings, intrauterine device/coil, double-barrier methods (e.g., sponge, spermicide, or condoms). Abstinence and/or vasectomized partner must agree to a second acceptable method of birth control (double-barrier) should the subject become sexually active.
    2. 2. A female is considered of non-childbearing potential if she is: postmenopausal (no menses for at least 12 months), without a uterus (hysterectomy) and/or both ovaries (oophorectomy), or bilateral tubal ligation.

Exclusion Criteria:

1. The presence of severe facial skin aging (as defined by Modified Griffiths' Scale, with an average score of 7-9) or minimal facial skin aging (as defined by Modified Griffiths' Scale, with an average score of 0-3).
2. Females who are pregnant, planning a pregnancy, or currently breast feeding during the study.
3. Any uncontrolled systemic disease.
4. History of autoimmune connective tissue disease.
5. Current use of immunosuppressive medication.
6. Weight change of greater than 10% during the study period.
7. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
8. Active dermatitis (including but not limited to atopic dermatitis, psoriasis, rosacea, acne, melasma, etc.), active infections, or other skin condition in the proposed treatment area that in the investigator's opinion might interfere with the evaluation of study parameters.
9. Mesotherapy; dermal fillers, biostimulator injectables; radiofrequency device treatments; microfocused ultrasound device treatments; laser and light-based device treatments; microneedling; cryolipolysis; high intensity focused electromagnetic energy device treatment; or surgery during the 12-month period before study treatment. Botulinum toxin injections (Botox, Dysport, Xeomin, Daxify, Jeuveau) during the 6-month period before study treatment.
10. Any investigational treatment for skin quality of the cheeks during the 12-month period before the study treatment.
11. Creams/cosmeceuticals and/or home therapies for the prevention or treatment of skin fine lines, wrinkles, radiance, elasticity, firmness, or smoothness in the treatment area during the 4-week period before study treatment and throughout the course of the study.
12. Subjects with scarring in the treatment areas. Subjects with a history of keloids will be excluded.
13. Subjects who spray tanned or used sunless tanners in the treatment areas 4 weeks prior to study treatment.
14. History of bleeding disorder, concomitant use of anticoagulants, history of connective tissue disease (e.g., lupus, scleroderma), history of Bell's Palsy, epilepsy, smoking, and/or current pregnancy or breastfeeding.
15. Inability to ambulate following the procedure.
16. History of lidocaine and/or tetracaine sensitivity deemed by the investigator to preclude subject from enrolling into study.
17. Individuals with known allergies or sensitivities to any of the ingredients of any topical or injectable products being used in this study.
18. Subjects planning any cosmetic procedure to the treatment area during the study period, other than the treatment that will be performed by the investigator.
19. Use of topical steroids, retinoids/retinols, or vitamin C to the face within the previous 2-weeks of screening.
20. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female at birth
Enrollment: 24 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Global Fine Lines | Screening, Day 30, Day 60
  Score 0 no fine lines thru 9 numerous, many fine lines
Overall Hyperpigmentation | Screening, Day 30, Day 60
  Score 0= no hyperpigmentation thru 9= significant hyperpigmentation
Skin Tone Evenness | Screening, Day 30, Day 60
  Score 0= Very even tone thru Score 9= Uneven, discolored appearance (brown and/or red colors)
Skin Firmness | Screening, Day 30, Day 60
  Score 0= Firm, tight feeling skin thru Score 9= Loose, lax feeling skin
Skin Radiance/ Brightness | Screening, Day 30, Day 60
  Score 0= Very radiant, luminous or glowing appearance thru Score 9= Very dull/ matte and/or sallow skin appearance
Skin Texture Smoothness | Screening, Day 30, Day 60
  Score 0= Very smooth, even-looking skin texture, no roughness thru Score 9= Very rough, pronounced, extensive visible skin roughness
Global Wrinkles | Screening, Day 30, Day 60
  Score 0= No wrinkles present, no visible deep, wide and long wrinkles, skin looks smooth thru Score 9= Numerous wrinkles, deep, wide and long, densely packed together in the treatment area

SECONDARY OUTCOMES:
Physical Global Aesthetic Improvement Scale | Day 30 and Day 60
  Assess improvement of Abdominal skin laxity:
  Much Improved 2 Improved 1 No Change 0 Worse -1 Much Worse -2
Subject Global Aesthetic Improvement Scale | Day 30 and Day 60
  Assess improvement of Abdominal skin laxity:
  Much Improved 2 Improved 1 No Change 0 Worse -1 Much Worse -2

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center, San Diego, California, United States